CLINICAL TRIAL: NCT01821469
Title: Functional Correlates of Bipolar Disorders and Effects of the Psychoeducation. Assessment by Functional and Anatomic Neuroimaging.
Brief Title: Functional Correlates of Bipolar Disorders and Effects of the Psychoeducation. an fMRI Study
Acronym: BIP-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, AdministrateurDRC, Professor, University Hospital, Grenoble
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EssaiClinique_"BIP-ED"; 2011-A00425-36 (Other: ID RCB)
Record Dates: First submitted 2012-11-06; First posted 2013-04-01 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Conditions Influencing Health Status; Bipolar Disorders
Keywords: bipolar disorders; euthymic; psychotherapy; Functional magnetic resonance imaging
MeSH Terms: conditions — Bipolar Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- psychoeducation (Experimental): psychoeducation (12 weeks)
  Interventions: Behavioral: psychoeducation

INTERVENTIONS:
Behavioral: psychoeducation — Bipolar disorders are educated to learn about their pathology

SUMMARY:
This research project follows two main objectives: 1) Assess anatomical and functional cerebral abnormalities in bipolar disorder. 2) Evaluate anatomical and functional changes after the application of a psychoeducational program in these patients. Specifically, this project aims to assess neurophysiological (fMRI - activation and functional connectivity) and neuroanatomical (morphometry and diffusion tensor imaging) specificities related to bipolar disorders and the therapeutic response to the psychoeducation. The results of this thesis project would also contribute to the validation of a pathophysiological model of the bipolar disorder.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of bipolar disorders
* euthymic (Montgomery and Asberg depression rating scale < 10, Young Mania rating scale < 10)

Exclusion Criteria:

* other concomitant psychiatric disorders

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-05; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
fMRI measurement (neurophysiological [fMRI - activation and functional connectivity]) | measurements were performed at T1 and T2 (up to 3 months)
  measurements were performed before (T1) and after (T2) educational program of 12 sessions .One session last one hour and half once a week (they come at the hospital for all sessions : i.e. during 12 weeks). Thus, T1 to T2 is 3 months (average).

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Bougerol, professor, Principal Investigator — CHU grenoble pôle psychiatrie et neurologie
Locations (1):
- Ums Irmage, Grenoble, France

REFERENCES:
- [Derived] Favre P, Polosan M, Pichat C, Bougerol T, Baciu M. Cerebral Correlates of Abnormal Emotion Conflict Processing in Euthymic Bipolar Patients: A Functional MRI Study. PLoS One. 2015 Aug 5;10(8):e0134961. doi: 10.1371/journal.pone.0134961. eCollection 2015. PMID 26244883